CLINICAL TRIAL: NCT00236535
Title: A Comparison of the Efficacy and Safety of Tramadol HCl/Acetaminophen Versus Hydrocodone Bitartrate/Acetaminophen Versus Placebo in Subjects With Acute Musculoskeletal Pain
Brief Title: A Study of the Efficacy and Safety of Tramadol HCl/Acetaminophen, Hydrocodone Bitartrate/Acetaminophen and Placebo in Patients With Pain From an Ankle Sprain With a Partial Torn Ligament
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002815
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Sprains and Strains; Pain
Keywords: musculoskeletal; Pain; sprained ankle; ligament; sprain; ankle
MeSH Terms: conditions — Sprains and Strains; Pain; Ankle Injuries | interventions — Tramadol; Acetaminophen; Hydrocodone

INTERVENTIONS:
Drug: tramadol HCl + acetaminophen; hydrocodone bitartrate + acetaminophen; placebo

SUMMARY:
The purpose of this study is to explore the pain-relieving effects and safety of two analgesic treatment regimens as compared to placebo in patients experiencing acute musculoskeletal pain. Patients who are experiencing at least moderate acute musculoskeletal pain from an ankle sprain severe enough to require prescription pain relief medication will be randomized to receive either tramadol HCl/acetaminophen, hydrocodone bitartrate/acetaminophen or placebo.

DETAILED DESCRIPTION:
Tramadol HCl/acetaminophen is approved for short-term (five days or less) management of acute pain. The combination of tramadol HCl/acetaminophen provides a more rapid onset of action compared with tramadol HCl alone and a longer duration of action than acetaminophen alone. Therefore, the combination of tramadol HCl/acetaminophen may be effective for the treatment of acute musculoskeletal pain. The current study is a multicenter, randomized, double-blind, inpatient/outpatient, active-controlled, placebo-controlled, parallel-group study. Patients who are experiencing at least moderate acute musculoskeletal pain from an ankle sprain severe enough to require prescription medication will be enrolled. Patients will be randomized to receive either oral tramadol HCl/acetaminophen, hydrocodone bitartrate/acetaminophen or placebo. Patients will receive 2 capsules tramadol HCl/acetaminophen 37.5/325 milligrams or 1 capsule hydrocodone bitartrate/acetaminophen 7.5/650 milligrams + 1 capsule placebo or 2 capsules placebo. Patient may take 1 or 2 capsules up to 4 times daily as needed but no more than 8 capsules per day for 5 daysThe first dose of study medication will be given at the study site. Patients will complete a Pain Visual Analog Scale, Pain Relief Rating Scale and Pain Intensity Scale at 1, 2, 3 and 4 hours after the first dose of study medication. On Day 1, after the 4-hour evaluations, patients will be dispensed study medication for use throughout the rest of the study. Patients will also evaluate and record in a daily diary the pain intensity ratings and pain relief scores for Days 1-5 of the double-blind phase. At the final visit, patients will complete a Pain Intensity Scale and Pain Relief Rating Scale, an Activity Impairment Assessment and a Subject Overall Medication Assessment. At the first dose, patients are dispensed 2 capsules of study medication. Thereafter, patients may take 1 or 2 capsules of study medication orally up to 4 times per day, as needed for pain, but no more than 8 capsules per day. The objective of this study is to compare the pain-relieving effectiveness and safety of tramadol HCl/acetaminophen versus hydrocodone bitartrate/acetaminophen versus placebo for the treatment of acute musculoskeletal pain from an ankle sprain with a partial ligament tear.

2 capsules tramadol HCl/acetaminophen 37.5/325 milligrams or 1 capsule hydrocodone bitartrate/acetaminophen 7.5/650 milligrams + 1 capsule placebo or 2 capsules placebo; patient may take 1 or 2 capsules orally up to 4 times daily as needed but no more than 8 capsules per day for 5 days

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute ankle sprain with a partial ligament tear within 48 hours of study entry
* At least moderate pain from the ankle sprain at baseline and before first dose of study medication
* In generally good health
* If female of childbearing potential, using acceptable method of birth control

Exclusion Criteria:

* Use of ibuprofen within 6 hours or topical pain relievers within 12 hours of study entry
* Use of tramadol HCl, tramadol HCl/acetaminophen, or hydrocodone bitartrate/acetaminophen within 30 days of study entry
* Use of epilepsy or antidepressant medications 3 weeks before the study entry
* Chronic use of pain medications or muscle relaxants for any reason during the study
* No use of steroid medications (oral or inhaled) on a chronic basis
* Required hospitalization to treat the ankle sprain
* Head trauma
* Pain greater than the pain caused by the ankle sprain
* Complete ligament tear
* Bone fractures on x-ray
* Required physical therapy, other than for crutch training
* History of kidney damage
* Pregnant or breast-feeding patients
* Condition that might affect the way the body absorbs or processes the study medication
* Major psychiatric disorder, history of attempted suicides/suicidal tendencies
* History of substance abuse or chronic alcohol abuse in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2003-12; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Total pain relief (TOTPAR) over 4 hours on Day 1 after the administration of the first dose of study medication

SECONDARY OUTCOMES:
Sum of Pain Intensity Differences; Sum of Pain Relief Intensity Differences; Pain Visual Analog Scores; mean daily pain intensity and relief; final pain intensity, relief and activity impairment assessment; subject overall medication assessment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Hewitt DJ, Todd KH, Xiang J, Jordan DM, Rosenthal NR; CAPSS-216 Study Investigators. Tramadol/acetaminophen or hydrocodone/acetaminophen for the treatment of ankle sprain: a randomized, placebo-controlled trial. Ann Emerg Med. 2007 Apr;49(4):468-80, 480.e1-2. doi: 10.1016/j.annemergmed.2006.08.030. Epub 2006 Nov 20. PMID 17113683
- See also: A Comparison of the Efficacy and Safety of Tramadol HCl / Acetaminophen Versus Hydrocodone Bitartrate / Acetaminophen Versus Placebo in Subjects with Acute Musculoskeletal Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=491&filename=CR002815_CSR.pdf